CLINICAL TRIAL: NCT06163105
Title: The Effect of Gland Expression on the Regeneration of Meibomian Gland
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ngoc Van Anh Le, MD, Principal Investigator, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0868/66
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Meibomian Gland Dysfunction
Keywords: Meibomian gland expression; squeezing; Regeneration; Morphology
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meibomian gland expression (MGX) (Experimental): * In-office MGX every 2 weeks
  * Lid hygiene at home once daily for 12 weeks
  * Preservative-free artificial tears (0.18% sodium hyaluronate) 4 times daily for 12 weeks
  Interventions: Procedure: Meibomian gland expression (MGX)
- Control group (No Intervention): * Lid hygiene at home once daily for 12 weeks
  * Preservative-free artificial tears (0.18% sodium hyaluronate) 4 times daily for 12 weeks

INTERVENTIONS:
Procedure: Meibomian gland expression (MGX) — The MGX procedure has a standardized protocol in lid spa at Chula's Refractive Surgery Center every 2 weeks (totally 6 sessions). During the study, all MGX procedures will be conducted by the same nurse following these steps:
  1. Topical anesthesia by Tetracaine 0.5%
  2. Clean the eyelids by gauzes with commercial available foam
  3. Warm the eyelids by Blephasteam machine for 10 minutes
  4. Instill Tetracaine 0.5% again
  5. Use Mastrota paddle and Q-tip to squeeze the gland
  6. Clean the lid margin by commercial available foam
  7. Use Moxifloxacin 0.5% eyedrop
  Other Names: Meibomian gland squeezing
  Arms: Meibomian gland expression (MGX)

SUMMARY:
The goal of this clinical trial is to compare the percentage of meibomian gland (MG) dropout in patients who are treated with additional meibomian gland expression (MGX) and in patients who are not. The main question[s] it aims to answer are:

* Does additional MGX reverse MG dropout and support regeneration of MG?
* Does additional MGX have better effect on tear film stability, MG function, lid morphology, tear cytokines than lid hygiene alone?

Methods:

Participants will be randomly assigned into MGX group as a treatment group and control group to assess study outcomes. The basic treatment of the 2 groups included lid hygiene once daily and artificial tear. The treatment duration lasts for 12 weeks. Patients will be examined at baseline, at 4-week, 8-week, 12-week visit for MG dropout percentage, MG morphology, lid margin abnormalities, Meibum assessment, tear film, tear cytokines and pain score to see if additional MGX can regenerate MG better than lid hygiene alone.

DETAILED DESCRIPTION:
1. Study design: an assessor-blinded, randomized, controlled trial
2. Target population: MGD patients having mild to moderate MG dropout from Out-clinic at King Chulalongkorn Memorial Hospital (KCMH).

4) Randomization and blinding Permuted block randomization will be used. After recruiting in this study, participants who meet the eligibility criteria will be divided into 2 groups by research assistant. There is an independent ophthalmologist (A.L) who is blinded to treatment allocation.

5)Data collection Demographic characteristics, numeric rating scale-11 (NRS-11) and ocular surface disease index (OSDI) will be collected by interviewing. Other parameters will be collected by slit lamp examination, specific machines or further investigations. All the data will be filled in the medical record. The participants will be identified on medical record by a unique research number, not by name or identification (ID) number (apart from on the consent form and enrollment log). Patient's ID, name, surname, and phone number will be stored in different file by the research assistant. The data will be locked up and destroyed 5 years after the study ends.

When the patients are recruited in the study, the patients will be provided information sheet and explained about the study. If the patients agree to participate in the study, they will be asked to sign the consent form. Then, they will be appointed to return to the Refractive Surgery Center in the next day for examination and tear collection between 1 pm to 3 pm because some cytokines are independent diurnal rhythms.

All outcome data will be collected by one single masked investigator (A.L). The data will be collected at 4 time points (day 0, week 4, week 8 and week 12). At baseline and 12-week post treatment, participants are required to be at the hospital on time within the period of 1 pm to 3 pm for tear collection. In each visit, the examination must be done in correct order in order not to avoid the results of outcomes. These steps include:

* Tear collection
* Evaluating the ocular symptoms
* Measuring lipid layer thickness
* Slit-lamp examination (tear break up time, lid margin abnormality, meibum expressibility and meibum quality)
* Non-contact infrared Meibography
* Evaluating adverse events

  8) Sample size: There is no previous study showing the difference in Meibomian gland dropout area between these groups. Our expert's opinion about minimal clinical difference is 10%. The standard deviation of meibomian gland dropout area in obstruction MGD patients is 16.7%. We use the formula for a trial with an equal allocation ratio and repeated measurements. This will be inflated for a 10% drop out, giving a total sample size of 32 per group (total sample size of 64).
* Statistical analysis:

Stata (version 17) software are utilized. All statistical analyses were undertaken by a researcher who are blinded to group allocation. The data were analyzed using an intention-to-treat (ITT) framework, which included all participants randomized in the study, regardless of the treatment type or exposure received. Per protocol (PP) is added as a supportive analysis. PP analysis will exclude the participants who do the lid hygiene less than 20 days per month or using any other treatment than advice. A significance level of 5% was used in all statistical tests.

Demographic data will be interpreted by descriptive analysis. The primary outcome is the change in meibomian gland percentages of each eyelid from baseline over all follow-up visits analyzing by linear mixed models with random intercept for patient, adjusting for baseline Meibomian gland percentage in the study participants and modelling time as a discrete variable. Marginal models will be used to predict the discrete changes at each study month. OSDI, tear break up time and lipid layer thickness are analyzed by linear mixed models (LMM). Lid abnormalities, meibum score and MG morphology will be analyzed by generalized linear mixed model (GLMM). Cytokine levels will be analyzed by unpaired t test.

9) Missing data management: If a patient chooses to withdraw from the study, the reason for withdrawal will be documented. These reasons will be valuable for analyzing the results later on. Multiple imputation method will be used to handle with missing data.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of obstructive MGD
* Visible Meibomian gland dropout of upper and lower eyelid from grade 1 to grade 2 (Arita's meiboscale)
* If both eyes meet above criteria, only right eye is chosen

Exclusion Criteria:

* Diagnosis with secondary MGD
* Having any eyedrop other than eye lubricant within the last 3 months
* Any kind of eyelid treatment related to MGD within the last 6 months
* History of ocular trauma, ocular surface surgery or eyelid surgery
* History of intraocular surgery less than 6 months
* Eyelid botulinum toxin injection within the last 6 months
* Ocular diseases other than dry eye
* Pregnant or breast-feeding
* Wearing contact lens
* Using any hormones therapy, anti-inflammatory drugs, tetracycline and macrolides
* Refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Meibomian gland dropout percentage | Baseline, week 4, week 8, week 12
  The dropout percentage of upper and lower eyelid is calculated by (Area of Meibomian gland dropout) / (Area of tarsal plate)*100%. Non-contact infrared Meibography is carried out using Oculus Keratograph 5M with upper and lower eyelids everted consecutively. To calculate the dropout area percentage of each eyelid, the investigator analyzes the images by utilizing the ImageJ software.

SECONDARY OUTCOMES:
Meibomian gland morphology | Baseline, week 4, week 8, week 12
  Meibomian gland morphology includes:
  * Distorted glands: glands not parallel to normal glands with torsion ≤45°
  * Tortuous glands: glands not parallel to normal glands with torsion >45°
  * Hooked glands: glands curling back at the distal end
  * Overlapping glands These variables are binary variables (Yes/No) They are analyzed by meibography images taken by Keratograph 5M
Lipid layer thickness | Baseline, week 4, week 8, week 12
  Lipid layer thickness measurement by Lipiview interferometer. For each eye, a 20-second video will be recorded to quantify the thickness of tear film's lipid layer in interferometric color unit (ICU) which corresponds to 1 nanometer. Images are captured while the participant focuses on the internal target. They are allowed to blink naturally during this process. Patients should not use any artificial tear for at least 4 hours and should not use ointments for at least 24 hours prior to LipiView assessment.
Lid margin abnormality | Baseline, week 4, week 8, week 12
  Lid margin abnormality score in upper and lower eyelid will be calculated by summing the score of 4 aspects:
  * Telangiectasia (0: No or slight redness in lid margin conjunctiva and no telangiectasia, 1: Redness in lid margin conjunctiva and no telangiectasia crossing meibomian gland orifices, 2: conjunctival redness and telangiectasia < 1/2 full length of the lid, 3: conjunctival redness and telangiectasia ≥ 1/2 full length of the lid)
  * Plugging (0: No plugging, 1: < 3 plugging, 2: ≥3 plugging with a distribution of <1/2 full length of the lid, 3: ≥3 plugging with a distribution of ≥ 1/2 full length of the lid)
  * Thickening (0: No thickening, 1: Lid margin thickening with or without localized rounding, 2: diffuse rounding)
  * Irregularity (0: No irregularity, 1: <3 lid margin irregularities with shallow notching, 2: ≥3 lid margin irregularities or deep notching)
Meibum quality | Baseline, week 4, week 8, week 12
  The meibum quality score was conducted by Evaluator (TearScience). Meibum quality score is obtained by evaluate each of eight glands of the central third of the lower eyelid on a scale of 0 to 3 for each gland (0: clear, 1: cloudy, 2: Cloudy with debris (granular), 3: Thick, like toothpaste). Total score ranges from 0 to 24.
Meibum expressibility | Baseline, week 4, week 8, week 12
  The meibum expressibility score was conducted by Evaluator (TearScience). Meibum expressibility is evaluated on a scale ranging from 0 to 3 for five glands of the lower eyelid. The assessment is based on the number of glands that can be expressed.
  0: All glands, 1: 3-4 glands, 2: 1-2 glands, 3: no gland
Pain level | Baseline, week 2, week 4, week 6, week 8, week 10
  MGX group is assessed pain level by interview the patients within 15 minutes after the procedure by a numeric rating scale-11 (NRS-11). Pain levels ranges from 0 to 10 as follows: 0, no pain; 10, worst possible pain; 1 to 3, mild pain; 4 to 6, moderate pain; and 7 to 10, severe pain
Adverse events | week 4, week 8 and week 12
  Adverse events will be questioned and recorded after the MGX and in every follow-up visit (week 4, week 8 and week 12) in both 2 groups. The examination using slit-lamp biomicroscopy to examine the eyelashes, eyelids, conjunctiva, cornea, anterior chamber, and lens is performed to detect any adverse events such as conjunctival congestion and eyelid puffiness, subconjunctival/lid hemorrhages, chalazion, acute conjunctivitis and keratitis.

CONTACTS AND LOCATIONS:
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand